CLINICAL TRIAL: NCT04788992
Title: Evaluation of a Dementia Care Training With Virtual Reality and Support Program for Home Care Staff
Brief Title: Dementia Care Training With Virtual Reality and Support for Home Care Staff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tzu Chi University (Other)
Responsible Party: Principal Investigator, Huei-Chuan Sung, Associate professor, Tzu Chi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: YLH-IRB-10815
Record Dates: First submitted 2021-03-02; First posted 2021-03-09 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Dementia
Keywords: Home care staff; dementia care; virtual reality
MeSH Terms: conditions — Dementia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: two-group cluster randomised controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): receive dementia care training
  Interventions: Other: Intervention group
- Control group (Active Comparator): receive dementia care training without virtual reality activity
  Interventions: Other: Control group

INTERVENTIONS:
Other: Intervention group — Dementia care training consists of dementia care e-books, dementia virtual reality activity and peer support program.
  Arms: Intervention group
Other: Control group — Dementia care training consists of dementia care e-books and peer support program without dementia virtual reality activity
  Arms: Control group

SUMMARY:
This study aims to evaluate a dementia care training with virtual reality and peer support program on dementia care knowledge, attitude, care competence, work stress, and empathy of home care staff.

DETAILED DESCRIPTION:
Home care staff often have insufficient knowledge and skills of caring people with dementia at home. Many lack empathy for those with dementia. Training courses for home care staff often are not developed according to their educational background and workplace needs.

This two-group cluster randomised controlled trial aims to evaluate a dementia care training with virtual reality and peer support program on dementia care knowledge, attitude, care competence, work stress, and empathy of home care staff.

The dementia care training consists of dementia care e-books, dementia virtual reality activity and peer support program.

The interventional group will receive a dementia care training using dementia care e-books, dementia virtual reality activity and peer support program.

The control group will only receive dementia care e-books and peer support with no dementia virtual reality activity.

Both groups will be assessed for their dementia care knowledge, attitudes, care competence, work stress and empathy at baseline, month 3, and 6.

ELIGIBILITY:
Inclusion Criteria:

* age 20 to 65 years
* Taiwanese nationality
* had worked as a home care staff for at least three months
* had experience in providing home care for patients with dementia
* had a mobile phone or tablet and regular access to the internet

Exclusion Criteria:

* Home care staff who do not meet the inclusion criteria
* can not provide informed consent.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Dementia Knowledge Assessment Scale | 6 months
  To evaluate care staff's knowledge of dementia, range from 0-50
Approach to Dementia Questionnaire | 6 moths
  To evaluate care staff's attitude toward Dementia, range from 19-95
Sense of Competence in Dementia Care Staff Scale | 6 months
  To evaluate care staff's competence of caring for people with dementia, range from 16-68
Jefferson Scale of Empathy | 6 months
  To evaluate care staff's level of empathy toward patients, score range from 20-140

SECONDARY OUTCOMES:
Simple Work Stress Scale | 6 moths
  To evaluate level of work stress of care staff

CONTACTS AND LOCATIONS:
Overall Officials: Huei-Chuan Sung, PhD, Principal Investigator — Tzu Chi University
Locations (1):
- Mennonite Social Welfare foundation, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No